CLINICAL TRIAL: NCT04941547
Title: Association Between Cancer and Anti-synthetase Syndrome : a Multicenter Study
Brief Title: Association Between Cancer and Anti-synthetase Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Centre Hospitalier Universitaire Dijon (Other); CHU de Reims (Other); University Hospital, Strasbourg, France (Other); Hopitaux Prives de Metz, Groupe UNEOS (Other); Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2021PI055
Record Dates: First submitted 2021-06-22; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-05

CONDITIONS: Antisynthetase Syndrome
Keywords: cancer; idiopathic inflammatory myopathies
MeSH Terms: conditions — Antisynthetase syndrome; Neoplasms; Myositis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Among Idiopathic inflammatory myopathies, antisynthetase syndrome is meant to be rarely associated with cancer. However, clinical evidences of the association of those diseases led to the hypothesis that previous studies might have underestimated the prevalence of cancer in patients with antisynthetase syndrome. The aim of this study was to assess the prevalence of cancer in patients with antisynthetases syndrome in Grand Est and Bourgogne Franche-Comté regions.

DETAILED DESCRIPTION:
Idiopathic inflammatory myopathies area heterogeneous group of disease involving mainly muscles, which paraneoplastic feature has been well characterized, specifically in some subgroups such as dermatomyositis. In contrast, antisynthetase syndrome is thought to be rarely associated with cancer. However, clinical observations of the association of those diseases led us to the hypothesis that previous studies might have underestimated the prevalence of cancer in patients with antisynthetase syndrome. The aim of this study was to assess the prevalence of cancer in patients with antisynthetases syndrome in Grand Est and Bourgogne Franche-Comté regions, describing the type of cancer observed as well as clinical features of patients and diagnostic work-up leading to the diagnosis of cancer.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* positive antisynthetase antibodies (JO-1,PL12, PL17, EJ, OJ, KS, RS, YRS)

Exclusion Criteria:

* age under 18
* opposition to data collection
* no positive antisynthetase antibodies
* absence of clinical involvment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with antisynthetase syndrome, defined by the positivity of antisynthetase antibodies and the presence of at least one clinical involvment, are included, either with or without cancer, to allow comparison of patients according to the presence of cancer.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
cancer prevalence | baseline
  prevalence of cancer among patients with antisynthetase syndrome

SECONDARY OUTCOMES:
description of cancer type in patients with antisynthetase syndrome | baseline
  description of the type and stage of cancer in patients with antisynthetase syndrome
factors associated with cancer | baseline
  comparison of clinical and paraclinical features associated with cancer in patients with antisynthetase syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Moulinet, MD, Principal Investigator — CHRU de Nancy
Locations (1):
- Thomas Moulinet, Vandœuvre-lès-Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: No